CLINICAL TRIAL: NCT03326726
Title: Evaluation of the Area Covered by Medline 2% Chlorhexidine Gluconate Cloth Preoperative Skin Preparation
Brief Title: Evaluation 2% Chlorhexidine Gluconate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R16-034
Record Dates: First submitted 2017-10-23; First posted 2017-10-31 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Skin Coverage
MeSH Terms: interventions — Chromogranins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chlorhexidine Gluconate (Experimental): 2% CHG
  Interventions: Drug: 2% CHG

INTERVENTIONS:
Drug: 2% CHG — Chlorhexidine Gluconate
  Other Names: Medline 2% CHG cloth

SUMMARY:
Medline 2% CHG cloth (Active) - A single cloth from the pack was used per treatment area. The investigational test article was applied topically by vigorously scrubbing the skin in a back and forth motion for three minutes (and halfway through the 3-minute application time, the cloth was turned over) over the treatment area (7" x 10" of the subject's back), and the skin was allowed to air dry.

ELIGIBILITY:
Inclusion Criteria:

Healthy males of at least 18 years of age having skin within 6 inches of the test regions that were free of tattoos, dermatoses, abrasions, cuts, lesions or other skin disorders, with no history of sensitivity to CHG and were able to lie prone for up to 30 minutes.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Bashir, Principal Investigator — Microbac Laboratories, Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy males at least 18 years of age having skin within 6 inches of the test regions that were free of tattoos, dermatoses, abrasions, cuts, lesions or other skin disorders, with no histroy of sensitivity to CHG and able to lie prone for up to 30 minutes.
Groups:
- 2% CHG Cloth: 2% chlorhexidine gluconate cloth
Period: Overall Study
Arm/Group | 2% CHG Cloth
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 2% CHG Cloth
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethniticy: White | 7
  Race/Ethniticy: Black or African American | 7
  Race/Ethniticy: Hispanic or Latino | 2
  Race/Ethniticy: Asian | 11
  Race/Ethniticy: Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Medline 2% CHG Cloth Dosage of Coverage Area
Description: To measure the dosage of the coverage area of a single investigational test article, Medline 2% CHG cloth calculated in grams per square centimeter
Time Frame: 3 minutes
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | 2% CHG Cloth
Number analyzed (Participants) | 30
g/cm^2 | 0.0081 (0.0013)

2. Secondary Outcome: Post-application Drying Time
Description: To assess post-application drying time after a single dose topical application of Medline 2% CHG cloth. Drying time is defined as when the entire treatment area appears visibly dry.
Time Frame: Approximately 1 minute
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 2% CHG Cloth
Number analyzed (Participants) | 30
seconds | 70 (18)

ADVERSE EVENTS:
Time Frame: 3 days
Description: There were zero adverse events reported throughout the duration of the study.
Arm/Group | 2% CHG Cloth
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data remains confidential